CLINICAL TRIAL: NCT02098083
Title: Evaluation of Physical Therapy Interventions and Patient Characteristics on Functional Mobility Outcomes in Persons With Acute Stroke
Brief Title: Evaluation of Physical Therapy Interventions and Patient Characteristics on Outcomes
Acronym: PBE
Status: Withdrawn | Type: Observational
Why Stopped: Unable to collect data
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Karen McCain, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 092013-009
Record Dates: First submitted 2014-03-20; First posted 2014-03-27 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Acute Stroke
Keywords: acute; stroke; gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Data collection for this study will be done by clinicians working in inpatient rehabilitation units with persons with acute stroke. No interventions are included in this study. It is designed to capture trends in current clinical practice for persons with stroke. This data will be useful in identifying the most beneficial and effective walking treatments as well as most significant patient characteristics that impact recovery for persons acutely after stroke. All data collection will take place during the inpatient rehabilitation stay.

DETAILED DESCRIPTION:
All persons admitted to the inpatient rehabilitation unit will be screened for inclusion. Only those with a confirmed diagnosis of stroke (CVA) will be included. Data collection on the participants will begin at the time of admission and continue through discharge. Average length of stay for persons with stroke in inpatient rehabilitation units is 21 days. Some persons will stay fewer days and some will stay longer. Data collection will include key information on physical therapy interventions including gait training, balance training, group therapy, manual therapy, exercise, transfer training, stairs, family training, wheelchair training, modalities, discharge planning, seated and supine exercises. Other data will be collected including tone, motor control, sensation, gait endurance, falls, wounds, restraints, deep vein thrombosis, tracheostomy, feeding tubes and blood pressure. Additional data collection will include age, gender, race, length of time post stroke, time in rehabilitation, Functional Independence Measure scores, case mix group, discharge destination. In addition, physician history and physical as well as discharge summary will be collected, as will evaluation and discharge notes from therapies (physical, occupation, speech, social work). Patients will not be responsible for any costs associated with this data collection.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a confirmed primary diagnosis of stroke, within 6 weeks of onset, will be included.
* Persons will be between the ages of 16 and 80.
* Persons may have experienced a previous CVA if they experienced a full gait recovery.

Exclusion Criteria:

* Any patient with a history of stroke onset greater than 6 weeks prior to admission will not be included.
* In addition, persons with bilateral CVA will not be included as well as persons who were not ambulatory prior to the CVA.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons post stroke admitted to inpatient rehabilitation units
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
6-Minute Walk Test | Subjects will be followed for the duration of inpatient rehabilitation, an expected average of 4 weeks
  The 6-Minute Walk Test is a test of walking endurance that is valid and reliable for persons post stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Karen J McCain, PT, DPT, NCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (4):
- United States (4):
  - Baylor Institute for Rehabilitation, Dallas, Texas
  - Baylor All Saints, Fort Worth, Texas
  - Baylor Institute for Rehabilitation Frisco, Frisco, Texas
  - Baylor Medical Center of Irving, Irving, Texas